CLINICAL TRIAL: NCT03920774
Title: Natural History of Familial Dysautonomia
Brief Title: The Natural History of Familial Dysautonomia
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-01774
Record Dates: First submitted 2019-04-04; First posted 2019-04-19 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Familial Dysautonomia (Riley-Day Syndrome); Hereditary Sensory and Autonomic Neuropathies; Hereditary Sensory and Autonomic Neuropathy 3
MeSH Terms: conditions — Dysautonomia, Familial; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — optional blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Familial Dysautonomia: Patients diagnosed with familial dysautonomia, a genetic disorder that affects the development and survival of nerve cells in the autonomic nervous system. It primarily affects neurons that control involuntary actions like regulation of blood pressure and breathing. It also affects the sensory nervous system and the perception of pain, heat and cold.

SUMMARY:
The study will collect clinical information from patients with FD and allow them to give blood to help develop biological markers of the disease to aid diagnosis and treatment.

This is a non-invasive, non-interventional, observation study that poses only minimal risk for participants. The study will document the clinical features of patients with FD overtime by storing their routine clinical test results in a central database. The study will involve collaborators at other specialist clinics around the world who follow/evaluate patients with FD annually. Providing blood for future use is optional.

DETAILED DESCRIPTION:
Define the phenotypic characteristics, severity and clinical evolution of FD on a patient-by patient basis. Investigators will enroll patients with FD in a multi-center observational natural history study to evaluate their biochemical, neurological and autonomic phenotype. Investigators will follow patients to systematically study the onset and scaled severity of all clinical problems. Investigators will define progression rates of patients outside of a clinical trial to distinguish between static and progressive features, a challenge in congenital neuropathies. Investigators will continue banking blood to look for ways to monitor the disease phenotypes. Biomarkers that quantify renal, cardiovascular, respiratory, skeletal and cognitive aspects of the disease will be evaluated. This information is relevant when monitoring toxicity to drugs in clinical trials. Detailed clinical follow-up of patients with FD will allow investigators to determine when standard of care therapies (e.g., non-invasive ventilation, gastrostomy feedings) should be initiated and how these impact survival outcomes.

Specific Aim 2: Develop ways to measure progressive neurological deficits as outcome measures for future clinical trials. Investigators will test the hypothesis that worsening gait ataxia and progressive visual loss are caused by ongoing neuronal degeneration. Investigators will develop precise outcome measures based on these deficits to test the efficacy of new treatments. Investigators will prospectively evaluate longitudinal changes in the retinal structure (with optical coherence tomography) and visual function in a cohort of patients with FD. Investigators will determine the extent and severity of retinal abnormalities in all patients and how they change overtime. Investigators will establish whether structural abnormalities in the retina are correlated with disease severity and look for functional correlates as measured by visual acuity and color discrimination. Following the recent discovery that gait ataxia in patients with FD is the result of sensory deficits, investigators will perform quantitative assessments of passive joint angle matching at the knee to measure proprioceptive acuity. Investigators will determine how these measures change overtime as well as their impact on daily function and quality of life.

An organized, multi-site natural history study of patients with FD will enable investigators to define disease-specific outcomes for testing new therapies, a major breakthrough for these patients. The study also offers a unique opportunity to understand better how the brain develops when devoid of crucial sensory inputs.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age with a diagnosis of familial dysautonomia (FD) with molecular confirmation of the IKBKAP mutation.
* Ability to provide informed consent (or assent) and comply with the study protocol

Exclusion Criteria:

* Subjects that do not wish to be a part of the study.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will involve as many as 400 human subjects. Registered patients range from 3 months to 66-years in age. This is a natural history study that will collect information obtained as standard of care from patients with FD.
  The study will involve children as it is a genetic disease with onset at birth. Adult patients will also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-02-22 (Actual); Primary Completion 2027-02-21 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
1. To create a database of familial dysautonomia disorder that will serve as a phenotypic core | 5 years
  Investigators will create an enrollment database of patients with familial dysautonomia. All patients will have standardized phenotypic evaluations that will combine clinical, physiological and biochemical strategies to characterize complex autonomic phenotypes, both known and still undiscovered.

SECONDARY OUTCOMES:
To define the natural history of visual function and identify predictive biomarkers of disease progression and severity. | 5 years
  Investigators will map the natural history of visual function including retinal structure and visual acuity and test the hypothesis that worsening visual loss is caused by ongoing neuronal degeneration.
To define the natural history of gait ataxia and identify predictive biomarkers of disease progression and severity | 5 years
  Investigators will map the natural history of gait ataxia and test the hypothesis that progressive ataxia is correlated with increasing loss of proprioceptive acuity caused by ongoing death of sensory neurons.

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, MD, Principal Investigator — NYU Langone Health
Locations (2):
- Dysautonomia Center - School of Medicine -NYU Langone Medical Center, New York, New York, United States
- Sheba Medical Center - Safra Children's Hospital, Tel Litwinsky, Ramat Gan, Israel